CLINICAL TRIAL: NCT00795873
Title: OVATIO CRT and SITUS OTW LV Lead Post Approval Study
Status: Completed | Type: Observational
Sponsor: ELA Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ITAC07
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2012-03

CONDITIONS: Heart Failure
Keywords: Heart failure; cardiac resynchronization therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Post approval study measuring safety outcomes on the Ovatio CRT-D and SITUS OTW LV lead over 5 years.

ELIGIBILITY:
Inclusion Criteria:

* NYHA Class III/IV
* Stable medical regimen
* QRS greater than or equal to 130 ms
* LVEF less than or equal to 35%

Exclusion Criteria:

* VT of transient or reversible causes
* Incessant VT
* Currently implanted with a lead positioned through the coronary sinus (unless it is the SITUS OTW LV lead)
* Cardiac revascularization or angioplasty within the last month
* Heart failure due to correctable valve disease
* Chronic, medially refractory AT
* Enrolled in another clinical study that may confound the results of this study
* Life expectancy less than 6 months
* Inability to understand the purpose of the study or refusal to cooperate
* Inability or refusal to provide informed consent
* Unavailable for scheduled follow-up with the implanting practice
* Sensitivity to 1 mg dexamethasone sodium phosphate
* Less than 18 years of age
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients needing CRT therapy
Sampling Method: Non-Probability Sample
Enrollment: 2260 (Estimated)
Dates: Start 2008-12

PRIMARY OUTCOMES:
SITUS OTW LV lead complication free rate | 5 years

SECONDARY OUTCOMES:
System complication free rate | 6 months

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Advanced Cardiac Specialists, Mesa, Arizona
  - Southwest Cardiovascular Associates, Mesa, Arizona
  - Cardiovascular Associates of Mesa, Mesa, Arizona
  - Cardiovascular Medical Group of Southern California, Beverly Hills, California
  - Center of Interventional Cardiology, Encino, California
  - Pacific Arrhythmia Service, La Mesa, California
  - Walter Kerwin, M.D., AMC, Los Angeles, California
  - Payam Robert Yashar, M.D. Inc., Los Angeles, California
  - Valley Regional Arrhythmia Center, Tarzana, California
  - High Desert Heart Institute Medical Corp., Victorville, California
  - Delaware Cardiovascular Associates, Wilmington, Delaware
  - Florida Institute for Cardiovascular Care, Hollywood, Florida
  - Electrophysiology Consultants of Florida, Miami Beach, Florida
  - Central Gerogia Heart Clinic, Macon, Georgia
  - Oschner Clinic Foundation, New Orleans, Louisiana
  - Primary Care Cardiology Research, Ayer, Massachusetts
  - Internal Medicine & Cardiology Associates of SE New England, PC, Fall River, Massachusetts
  - Clipper Cardiovascular Associates, Newburyport, Massachusetts
  - Jackson Cardiology Associates, P.A., Jackson, Mississippi
  - Atul Prakash, M.D., Clifton, New Jersey
  - Cross County Cardiology, Edgewater, New Jersey
  - Hudson Heart Group, PC, Guttenberg, New Jersey
  - Cardiovascular Associates of Mountainside, PA, Mountainside, New Jersey
  - Joaquim J Correia, MD LLC, Newark, New Jersey
  - NJ Heart, Newark, New Jersey
  - Divagno Cardiology, Rochelle Park, New Jersey
  - The Heartcare Center, Saddle Brook, New Jersey
  - Clinical Cardiovascular Specialists, Columbus, Ohio
  - Toledo Clinic Inc., Toledo, Ohio
  - Cardiovascular Consultants, Inc., Tulsa, Oklahoma
  - Cardiac Consultants, PC, Lancaster, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Midlands Cardiology Associates, Columbia, South Carolina